CLINICAL TRIAL: NCT07372027
Title: A Prospective Study on the Efficacy and Cost-Effectiveness of Modified Single-Needle Distal Return Cannulation for Long-Term Arteriovenous Fistula Care in Maintenance Hemodialysis Patients
Brief Title: Single-Needle Distal Return for Long-Term Arteriovenous Fistula Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Municipal Hospital of Anhui Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASZH-2024-CS-HD-SNC-01
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hemodialysis Access; Arteriovenous Fistula; Arteriovenous Fistula Cannulation; Vascular Access; Vascular Access Complication
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Needle Distal Return (Experimental)
  Interventions: Procedure: Single-Needle Distal Return (SNDR) Cannulation
- Standard Two-Needle AVF Cannulation (Active Comparator)
  Interventions: Procedure: Standard Two-Needle AVF Cannulation

INTERVENTIONS:
Procedure: Single-Needle Distal Return (SNDR) Cannulation — For each hemodialysis session, only a single needle is used to cannulate the arteriovenous fistula (AVF) to establish arterial blood inflow. The venous return is established by cannulating a superficial vein in the distal lower extremity (such as the dorsal foot vein or a tributary of the great saphenous vein), which is separate from the AVF. This approach aims to minimize repetitive trauma to the AVF segment itself.
  Arms: Single-Needle Distal Return
Procedure: Standard Two-Needle AVF Cannulation — For each hemodialysis session, the established standard of care is followed. This involves cannulating the arteriovenous fistula (AVF) with two separate needles: one placed proximally (or in the arterial segment) to establish blood inflow, and a second placed distally (or in the venous segment) to return dialyzed blood. This is the conventional method for maintenance hemodialysis via an AVF.
  Arms: Standard Two-Needle AVF Cannulation

SUMMARY:
Background:

For millions of people worldwide with kidney failure, a well-functioning vascular access, like an arteriovenous fistula (AVF), is essential for life-sustaining hemodialysis. However, the standard method requires puncturing the same AVF with two needles three times a week, which over time can damage the vessel, leading to scarring, narrowing, and frequent failures. These complications often require repeated surgical or minimally invasive procedures (reinterventions), causing significant pain, high medical costs, and exhaustion of the patient's limited blood vessels.

New Approach:

This study will evaluate a modified puncture technique called the Single-Needle Distal Return (SNDR) strategy for long-term AVF care. Instead of using two needles in the AVF, only one needle is placed in the AVF to draw blood. The cleaned blood is then returned to the body through a second needle placed in a superficial vein in the foot or lower leg. This approach aims to reduce trauma to the critical AVF.

Study Plan:

This is a clinical study conducted at the Blood Purification Center of Anhui Medical University Affiliated Suzhou Hospital. We plan to enroll approximately 50 adult hemodialysis patients who use an AVF and are willing to try the SNDR technique. For comparison, we will also observe data from a similar number of patients receiving standard two-needle AVF care during the same period.

The study will last about three years. We will closely monitor patients using the SNDR technique to assess:

Effectiveness: Whether dialysis remains adequate (measured by Kt/V).

Safety: Rates of complications (like bruising or infection), dialysis machine alarms, and venous pressure during treatment.

Practical Benefits: Whether it reduces the need for repair procedures (reinterventions) and hospitalizations related to the AVF.

Economic Impact: Changes in healthcare costs.

Patient Experience: Patient tolerance and comfort with the technique. We will also analyze the characteristics of patients who successfully use this technique long-term to help identify who might benefit most from it in the future.

Potential Significance:

If proven successful and safe for long-term use, the SNDR strategy could help protect a patient's precious AVF, potentially reducing painful procedures, lowering costs, slowing down the exhaustion of blood vessels, and improving the quality of life for people on long-term dialysis. The findings may also guide better planning for vascular access care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years).

Diagnosis of end-stage kidney disease (ESKD) requiring maintenance hemodialysis (three times per week).

Reliable use of a native arteriovenous fistula (AVF) as the primary vascular access for at least the past 3 months.

Willing and able to provide written informed consent to participate in the study.

Adequate superficial venous vasculature in at least one lower extremity (e.g., dorsal foot veins, saphenous tributaries) as assessed by clinical evaluation and/or bedside ultrasound, deemed suitable for cannulation as a venous return site.

For the experimental (SNDR) group: Expressed willingness to adopt the single-needle distal return cannulation strategy.

For the control group: Currently receiving and willing to continue standard two-needle AVF cannulation.

Exclusion Criteria:

* Active systemic infection or localized infection at the potential cannulation sites (AVF or lower extremity veins).

Known severe coagulation disorder or thrombocytopenia (platelet count < 50 × 10⁹/L) that would pose a high risk of bleeding complications from cannulation.

Severe peripheral arterial disease or venous insufficiency in the lower extremities that contraindicates venous cannulation or may compromise limb perfusion.

Unstable cardiovascular status (e.g., uncontrolled heart failure, severe arrhythmias) as determined by the treating nephrologist, which would increase the risk associated with any change in dialysis procedure.

Documented severe cognitive impairment, psychiatric illness, or any condition that would impair the ability to provide informed consent or adhere to the study protocol.

Life expectancy less than 12 months due to non-renal comorbid conditions (e.g., metastatic malignancy).

Currently pregnant or breastfeeding.

Participation in another interventional clinical trial that could confound the outcomes of this study.

Anatomical or pathological condition of the AVF (e.g., extreme depth, aneurysm with overlying skin compromise, complete thrombosis) that precludes safe single-needle cannulation, as judged by the study vascular access team.

Inability to comply with the scheduled study visits and follow-up assessments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-12-15 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in dialysis adequacy (single-pool Kt/V) from baseline to study completion. | From enrollment to the end of the 24-month follow-up period.
Annualized rate of access-related reinterventions (e.g., angioplasty, thrombectomy, surgical revision). | From enrollment to the end of the 24-month follow-up period.

SECONDARY OUTCOMES:
Total access-related healthcare costs per patient-year. | From enrollment to the end of the 24-month follow-up period.
Rate of hospitalizations primarily due to vascular access complications. | From enrollment to the end of the 24-month follow-up period.
Incidence of cannulation-related adverse events (e.g., hematoma, infection, severe bleeding). | Assessed at each hemodialysis session throughout the study, up to 24 months.
Proportion of hemodialysis sessions with significant machine alarms requiring staff intervention. | Assessed at each hemodialysis session throughout the study, up to 24 months.
Patient-reported tolerance and satisfaction assessed via a standardized questionnaire. | At 6 months, 12 months, and at study completion (24 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hospital Affiliated to Anhui Medical University, Suzhou, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes